CLINICAL TRIAL: NCT05538273
Title: Optimal Management and Timing of Removal of Urinary Catheter Following Pelvic Surgery by the Gynecologic Oncology Surgeon
Brief Title: Optimal Management of Urinary Catheter in Gyn Onc
Status: Withdrawn | Type: Observational
Why Stopped: Study not activated, staff left institution.
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Eav Lim, Site Director, Gynecology Oncology, WellSpan Health
Other Study IDs: 1946054-1
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Urinary Retention
Keywords: urinary retention; postoperative; urinary complications; pelvic surgery; hysterectomy; gynecologic oncology
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Minimal invasive surgery: removal of urinary catheter postoperatively
  Interventions: Other: Early removal of urinary catheter postoperatively; Other: Late removal of urinary catheter postoperatively
- Laparotomy: removal of urinary catheter postoperatively
  Interventions: Other: Early removal of urinary catheter postoperatively; Other: Late removal of urinary catheter postoperatively
- Simple surgery: removal of urinary catheter postoperatively
  Interventions: Other: Early removal of urinary catheter postoperatively; Other: Late removal of urinary catheter postoperatively
- Radical surgery: removal of urinary catheter postoperatively
  Interventions: Other: Early removal of urinary catheter postoperatively; Other: Late removal of urinary catheter postoperatively

INTERVENTIONS:
Other: Early removal of urinary catheter postoperatively — removal of urinary catheter less than 24 hours after surgery
Other: Late removal of urinary catheter postoperatively — removal of urinary catheter greater than 24 hours after surgery

SUMMARY:
This is a combined retrospective observational study that will collect data on urinary catheter removal of patients who underwent pelvic surgery by a gynecologic oncologist to assess timing safety and its implications in postoperative care.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* female gender
* undergoing pelvic surgery for benign or malignant indications by a gynecologic oncologist

Exclusion Criteria:

* Age less than 18 years of age at the time of surgery
* pregnant
* individual is a prisoner

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who meets the eligibility criteria, undergoing pelvic surgery by a gynecologic oncologist. Simple and radical procedures included.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Urinary retention rate after urinary catheter removal postoperatively | 30 days after surgery
  urinary retention rate will be measured as need for re-catheterization postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- WellSpan York Hospital, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No